CLINICAL TRIAL: NCT03706586
Title: Is the Use of Higher Versus Lower Oxygen Concentration Feasible in the Delivery Room: a Pilot Trial
Brief Title: The Hilo Pilot -Trial to Assess Feasibility
Acronym: HiLo-Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 00084090
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Premature Infant; Respiratory Distress Syndrome
Keywords: Delivery Room; Resuscitation
MeSH Terms: conditions — Premature Birth; Respiratory Distress Syndrome | interventions — Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: outcome assessed will be unaware of group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 30% group (Active Comparator): Infants in the 30 % group will remain in 30% oxygen (O2) until 5 min of age. At 5 min of age, the clinical team will assess oxygen saturation (SpO2). If SpO2 is <85%, O2 should be increased by 10-20% every 60 sec to achieve SpO2 of 85% or greater or a SpO2 of 90-95% at 10 min of age. If SpO2 are greater than 95% at or before 5 min of age, O2 should be decreased stepwise (every 60 sec) with an aim to maintain SpO2 of 85% or greater during 5-10 min of age or 90-95% at and beyond 10 min of age.
  Interventions: Procedure: 30% group
- 60% group (Experimental): Infants in the 60 % group will remain in 60% oxygen (O2) until 5 min of age. At 5 min of age, the clinical team will assess oxygen saturation (SpO2). If SpO2 is <85%, O2 should be increased by 10-20% every 60 sec to achieve SpO2 of 85% or greater or a SpO2 of 90-95% at 10 min of age. If SpO2 are greater than 95% at or before 5 min of age, O2 should be decreased stepwise (every 60 sec) with an aim to maintain SpO2 of 85% or greater during 5-10 min of age or 90-95% at and beyond 10 min of age.
  Interventions: Procedure: 60% group

INTERVENTIONS:
Procedure: 30% group — Infants in the 30 % group will remain in 30% oxygen (O2) until 5 min of age. At 5 min of age, the clinical team will assess oxygen saturation (SpO2). If SpO2 is <85%, O2 should be increased by 10-20% every 60 sec to achieve SpO2 of 85% or greater or a SpO2 of 90-95% at 10 min of age. If SpO2 are greater than 95% at or before 5 min of age, O2 should be decreased stepwise (every 60 sec) with an aim to maintain SpO2 of 85% or greater during 5-10 min of age or 90-95% at and beyond 10 min of age.
  Arms: 30% group
Procedure: 60% group — Infants in the 60 % group will remain in 60% oxygen (O2) until 5 min of age. At 5 min of age, the clinical team will assess oxygen saturation (SpO2). If SpO2 is <85%, O2 should be increased by 10-20% every 60 sec to achieve SpO2 of 85% or greater or a SpO2 of 90-95% at 10 min of age. If SpO2 are greater than 95% at or before 5 min of age, O2 should be decreased stepwise (every 60 sec) with an aim to maintain SpO2 of 85% or greater during 5-10 min of age or 90-95% at and beyond 10 min of age.
  Arms: 60% group

SUMMARY:
Preterm birth, or birth before 37 weeks' gestation, is increasingly common, occurring in 8% of pregnancies in Canada. Preterm birth is associated with many health complications, particularly when the birth happens before 29 weeks' gestation. At this gestational age, the lungs are not fully developed and it is not uncommon for infants to have problems breathing at the time of birth. One complication that can arise is when an infant stops breathing and needs to be resuscitated. When preterm babies need to be resuscitated doctors must take special care because of the small infant size and the immaturity of the brain and lungs. Oxygen is used to resuscitate babies who need it, but unfortunately there is disagreement about the best oxygen concentration to use. Oxygen concentration is important because both too much and too little oxygen can cause brain injury. Our research aims to fill this knowledge gap by participating in an international clinical trial to compare the effects of resuscitating babies less than 29 weeks' gestational age with either a low oxygen concentration or a high oxygen concentration. The oxygen concentrations have been selected using the best available knowledge. During the first 2 months of the clinical trial we will treat all babies less than 29 weeks' gestation who need resuscitation with the oxygen concentration we are randomly assigned. Then in the next 2 months, we will treat babies using the other oxygen concentration. After the trial, we will determine whether the babies resuscitated with low oxygen or those resuscitated with high oxygen have better survival and long-term health outcomes. Our research fills a critical knowledge gap in the care of extremely preterm babies and will impact their survival both here in Canada and internationally.

DETAILED DESCRIPTION:
Purpose: Over the last 10 years, recommendations regarding the ideal level of oxygen for resuscitation in preterm infants have changed from 100%, down to low levels of oxygen (<30%), up to moderate concentration (30-65%). In addition, in 2010, oxygen saturation targeting was recommended as standard of care and this contributed to a change in clinical practice as clinicians were more likely and comfortable to start resuscitation at either 21% (room air) or titrated levels of oxygen such as 30-40%. When the guidelines were again revised in 2015, the International Liaison Committee on Resuscitation (ILCOR) acknowledged that a critical knowledge gap continued to exist for the resuscitation of the preterm infants <37 weeks, highlighting the need to provide more concrete guidelines. This leaves clinicians in a challenging position. Despite the advances that have been achieved in perinatal and neonatal care, neonates are still vulnerable to the consequences of the oxidative effects from hyperoxia as well as the deleterious effects from hypoxia. A large, multi-centre international trial of sufficient sample size that is powered to look at safety outcomes such as mortality and adverse neurodevelopmental outcomes is required to provide the necessary evidenced to guide clinical practice with confidence.

Hypothesis: the null hypothesis for this study is that the incidence of mortality or abnormal neurodevelopmental outcomes at 18-24 months corrected age will be no different by using either higher initial oxygen concentration of 60% compared to using lower initial oxygen concentration of 30% for resuscitation of preterm infants of 23 0/7- 28 6/7 weeks gestation.

Justification:

The use of supplementary oxygen may be crucial, but also potentially detrimental to premature infants at birth. High oxygen levels may lead to organ damage through oxidative stress, while low oxygen levels may lead to increased mortality. Excess oxygen exposure during the early post-birth period is associated with many complications and morbidities of preterm birth. Preterm infants have lower levels of anti-oxidant pathways consistent with their expected fetal environment of low oxygen exposure. Excess of oxygen free-radicals in infants intrinsically deficient in enzymatic antioxidants and non-enzymatic antioxidants may contribute to these morbidities. Pulmonary oxygen toxicity, through the generation of reactive oxygen and nitrogen species in excess of antioxidant defenses, is believed to be a major contributor to the development of bronchopulmonary dysplasia (BPD). Using lower oxygen concentrations at birth results in decreased oxidative stress markers and a decrease risk of developing BPD compared to higher oxygen concentrations. Other organs that may be damaged by such oxidative stress include kidneys, myocardium and the retina.

There is equally growing evidence that using lower oxygen concentrations will lead to lower oxygen saturation levels and bradycardia, which may lead to increased rates of mortality in this vulnerable group of infants. An individual patient analysis of clinical trials reported that 46% of preterm infants resuscitated with initial low oxygen concentration did not reach SpO2 of 80% at 5 min. This was associated with increased risk of major intraventricular hemorrhage (IVH), and an almost five times higher risk of death in this vulnerable group of infants. These data provide a warning note for the use of higher vs. lower initial oxygen concentration during delivery room resuscitation. As we proceed in determining a safe range for resuscitation of ELBW/ELGA infants, it is highly likely that the optimum level of oxygen concentration is likely between the two extremes of 21% and 100%.

Objectives: To determine whether initial resuscitation of preterm neonates with 60% versus 30% oxygen in the delivery room is feasible.

Research Method/Procedures: This will be a cluster crossover design, unmasked randomized controlled trial (RCT) comparing two oxygen concentrations at initiation of resuscitation. Infants will be placed on the resuscitation table with the initial steps of resuscitation carried out as per standard of care at each centre which usually follows current resuscitation guidelines. All centres will make every effort to establish adequate lung expansion using CPAP or positive pressure ventilation as needed. Enrolled infants will have a pulse oximeter sensor placed on the right arm in the first minute of life. Their resuscitation will be initiated with an oxygen concentration of 30% or 60% depending on the randomization sequence at the centre at the given time. Infants in the 30 % group will remain in 30% oxygen until 5 min of age unless the infant's heart rate (HR) remains 100/min or less and does not show a tendency towards progressive increase before reaching 5 min of age or infant needs chest compression and/or epinephrine. No alteration in oxygen concentration will be made for an infant who is responding to resuscitation efforts with HR progressively increasing as minutes go by. At 5 min of age, the clinical team will assess oxygen saturation. If the saturation is less than 85%, oxygen should be increased by 10-20% every 60 sec to achieve saturations of 85% or greater or a saturation of 90-95% at 10 min of age. If saturations are greater than 95% at or before 5 min of age, oxygen should be decreased stepwise (every 60 sec) with an aim to maintain saturations of 85% or greater during 5-10 min of age or 90-95% at and beyond 10 min of age. The procedure for infants in the 60% group will be identical. The intervention duration for the trial will be the first 5 min after birth followed by initial monitoring/action for the next 5 min where titration in oxygen concentration will be made to achieve stability making a total of 10 min for study intervention. Titration of oxygen before 5 min after birth will only be made if the infant remains bradycardic (HR less than 100) and does not show a tendency towards a sustained increase in HR or if the oxygen saturation exceeds 95%. If the infant does not respond to ventilation with increasing HR in the first 5 min after birth, steps to ensure effective ventilation should be done before oxygen is titrated.

Plan for Data Analysis:

Data will be analysed as intention-to-treat. Data will be compared using Student's t-test for parametric and Mann-Whitney U test for nonparametric comparisons of continuous variables, and Fisher exact for categorical variables. The data will be presented as mean (standard deviation (SD)) for normally distributed continuous variables and median (interquartile range (IQR)) when the distribution will be skewed. P-values will be 2-sided and p<0.05 will be considered statistically significant. Statistical analyses will be performed with SPSS Statistics for Macintosh, Version 27.0 (Armonk, NY: IBM Corp).

ELIGIBILITY:
Inclusion Criteria:

• Infants born at 23 0/7 weeks to 28 6/7 weeks' gestational age who will receive full resuscitation and are without major congenital abnormalities

Exclusion Criteria:

* Infants who are outborn - initial resuscitation not performed at the study centre
* Infants who are not born within the eligible gestational age range- this trial is specific to preterm infants
* Infants who are born with a major congenital abnormality- congenital abnormalities may affect oxygenation or neurodevelopmental outcomes
* Infants who will not receive full resuscitation at birth- these infants will not receive resuscitation

Max Age: 10 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of 30% or 60% oxygen at birth | 10 Minutes after birth
  Titration oxygen during respiratory support at birth

CONTACTS AND LOCATIONS:
Overall Officials: Georg Schmolzer, Principal Investigator — University of Alberta
Locations (1):
- Royal Alexandra Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Law BHY, Asztalos E, Finer NN, Yaskina M, Vento M, Tarnow-Mordi W, Shah PS, Schmolzer GM. Higher versus Lower Oxygen Concentration during Respiratory Support in the Delivery Room in Extremely Preterm Infants: A Pilot Feasibility Study. Children (Basel). 2021 Oct 20;8(11):942. doi: 10.3390/children8110942. PMID 34828655